CLINICAL TRIAL: NCT02791425
Title: Wearable Brain Computer Interface (BCI) to Assist Communication in Mechanically Ventilated Patients the Intensive Care Unit (ICU)
Brief Title: Brain Computer Interface for Communication in Ventilated Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The developer of the BCI left the institution so the study could not continue
Sponsor: University of Michigan (Other)
Collaborators: Michigan Institute for Clinical and Health Research (MICHR) (Unknown)
Responsible Party: Principal Investigator, Venkatakrishna Rajajee, Clinical Associate Professor, Neurosurgery and Neurology Medical Director, Neurointensive Care, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00100788
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Mechanical Ventilation; Nonverbal Communication; Intratracheal Intubation; Critical Illness
Keywords: Brain-Computer Interface; Intratracheal intubation; Mechanical ventilation; Nonverbal communication; Critical illness; Electroencephalography; Visual Evoked Potential
MeSH Terms: conditions — Nonverbal Communication; Critical Illness | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Computer Interface (BCI) device (Experimental): The patient uses the Brain Computer Interface (BCI) device in the ICU for communication for 2 hours a day for 3 consecutive days. The patient then uses a communication picture board for 2 hours a day for 3 consecutive days on the same days that the BCI device is used for comparison.
  Interventions: Device: Brain Computer Interface (BCI) device; Other: Communication picture board

INTERVENTIONS:
Device: Brain Computer Interface (BCI) device — A BCI system to facilitate communication in intubated patients. Patients use the device in the ICU for communication for 2 hours a day for 3 consecutive days.
Other: Communication picture board — The patient then uses a communication picture board for 2 hours a day for 3 consecutive days on the same days that the BCI device is used for comparison.

SUMMARY:
Objectives:

Specific Aim 1: To demonstrate the feasibility of using a Steady State Visual Evoked Potential (SSVEP) based Brain Computer Interface (BCI) device to facilitate communication of common patient needs in alert mechanically ventilated patients in the Intensive Care Unit (ICU).

Specific Aim 2: To determine patient, family and bedside nurse satisfaction with communication using the BCI device and elicit open-ended feedback to guide future device improvements

Design:

Translational pilot study of a Steady State Visual Evoked Potential (SSVEP) based BCI system to facilitate communication in intubated patients, with sequential use of the BCI device and a picture board.

Selection of the primary self-identified primary patient need on the BCI device will be compared to the icon selected on the picture board (reference standard). A patient satisfaction survey will then be provided to the patient or a family member following use for 2 hours a day for 3 consecutive days.

Primary outcome: Accurate selection of the illustrative icon on the brain computer interface representing the physical or emotional need self-identified by the patient as being the most common trigger for communication with the bedside nurse during their admission.

Secondary outcome: Selection by patients or family of "agree" or "strongly agree" with the statement "The Brain computer interface device allowed me to communicate my needs to the bedside nurse adequately".

Intervention: Use of the brain computer device in the ICU for communication for 2 hours a day for 3 consecutive days

Control/ Comparator: Sequential use of a communication picture board for 2 hours a day for 3 consecutive days, on the same days that the BCI device is used Sample Size: 30 mechanically ventilated but alert patients in the Intensive Care Unit

DETAILED DESCRIPTION:
BACKGROUND

An inability to consistently and effectively communicate their most fundamental physical needs is a major problem for mechanically ventilated ICU patients. Patients rate about 40% of communication sessions as difficult and more than a third of communications about pain as unsuccessful. Nurses initiate about 86% of all communication exchanges as it is typically very difficult for a voiceless ICU patient to initiate communication. Patients in the ICU therefore commonly suffer unrecognized pain and discomfort, feelings of loss of control and insecurity, depersonalization, anxiety, sleep disturbances, fear and frustration. Caregivers also frequently report feeling anxious and frustrated in not being able to adequately assess the needs of their patients. This inability to communicate effectively can lead to the inappropriate use of sedatives and prolongation of time spent on the ventilator, which may then lead to increased ICU length of stay and costs. Furthermore, the inability to communicate with caregivers hampers the ability of critically ill patients to be active participants in their treatment and in decision-making, including decisions to withdraw or withhold life-sustaining treatment.

The use of picture boards with icons representing common patient needs and complaints (pain, fear, hot/ cold, thirst, bedpan etc) has been shown to improve nurse-patient communication for patients in the postoperative period on the ventilator. These picture boards are widely available in most ICUs and are the closest thing to a current standard for communication with voiceless mechanically ventilated patient, for the purposes of addressing fundamental physical and emotional needs. Recent pilot studies have described the use of computer-assisted communication using touch sensitive screens, eye blink detectors and gaze trackers to enable communication in the ICU patient. The majority of patients and hospital staff surveyed in these studies indicated that the use of a computer-assisted communication device improved the ability to respond to patient needs and address patient comfort. Gaze and eye blink tracker systems are expensive, however, while touch sensitive screens may not be suitable for the many ICU patients with weakness and restriction in motor ability. Patients in the ICU, particularly those with neurological illness, frequently suffer from significant weakness and loss of co-ordination, however, limiting their ability to use their arms and hands to indicate the appropriate item on the board. While patients in the neuroICU are frequently weak because of focal brain injury, about a quarter of patients requiring mechanical ventilation in other ICUs may have significant weakness from critical illness neuropathy and myopathy, limiting their ability to use their hands to select the appropriate icon on a picture board. There are several patient populations, however, for whom the use of a picture board or touch screen is impossible, including patients with high spinal cord injury, advanced ALS and brainstem stroke, who are voiceless, but also typically have no useful motor function of their limbs. These patients are "locked-in", to varying degrees, awake and alert but with no control of bodily function or ability to articulate and communicate using standard forms of communication.

The use of Brain Computer Interface (BCI) devices to facilitate communication in "voiceless" patients has recently generated interest. A BCI translates deliberate, voluntary modulation of cerebral electrical activity, typically recorded by electroencephalography (EEG) into computer commands. A variety of BCI devices have been used to permit patients with advanced Amyotrophic Lateral Sclerosis (ALS), high spinal cord injury and brainstem stroke with the locked-in-syndrome, who have no voluntary use of their limbs, to communicate to varying degrees. These devices have typically been evaluated in the rehabilitation setting, following the period of acute medical illness, or at home. No study has evaluated the use of a BCI device to assist with communication of the typical physical and emotional needs/ complaints of the critically ill. This is significant, not only for patients with spinal cord injury and stroke, most of who are initially admitted to an ICU, but to the potentially large number of ICU patients who cannot use a picture board or other finger contact system because of critical illness neuropathy/ myopathy or acute brain injury causing weakness. Our focus is on creating a steady state visual evoked potential (SSVEP) based, wireless BCI system to facilitate communication with intubated ICU patients., The wearable BCI device of interest in this study functions through visual attention to illustrative icons displayed on an electronic screen. The icon, which may depict a common ICU patient need, such the need for repositioning or common patient complaint, such as pain, can be displayed as a symbol. The patient can, thereby, communicate by looking at a specific item depicting their need or complaint. This wearable device is entirely noninvasive and without significant risk to patients, functioning only to record and translate EEG signals. The device will communicate wirelessly with the user interface (UI) that can be either a tablet or the flat screen TV monitor that is present in every ICU patient room. The proposed prototype provides a user interface that includes basic functions that are typically used in communication between nurses and patients in the ICU.

STUDY DESIGN

This is a translational pilot study of a Steady State Visual Evoked Potential (SSVEP) based BCI system to facilitate communication in intubated patients. After obtaining informed consent from the patient or their legally authorized representative, 30 patients will be recruited from the medical, surgical, cardiac, cardiothoracic and neurological intensive care units at the University of Michigan, Ann Arbor over a period of 12 months. Approval has been obtained from the Institutional Review Board of the University of Michigan (HUM00095052).

Screening for delirium and ability to participate in the study:

Potential subjects will be identified by members of the primary ICU team, who will then contact a study investigator. Subjects will need to be off all sedating medicines with return to full wakefulness prior to further evaluation. Patients meeting the above eligibility criteria who consent to participate in the study will then undergo further testing by an investigator to confirm that the patient is sufficiently alert and attentive to communicate AND is capable of consistently selecting items through volitional finger contact. The patient will then undergo a screening evaluation with the BCI device to confirm that their individual EEG signal can be detected and interpreted by the device.

Patient complaints/ needs: The investigators will evaluate the ability of subjects to accurately select a specific need or complaint from 10 common needs/ complaints.

1. "I am in pain"
2. "I have difficulty breathing"
3. "I need to be suctioned"
4. "I need to have a bowel movement"
5. "I need to pee/ pass urine"
6. "I am thirsty"
7. "I am hungry"
8. "I need to have my position in bed changed"
9. "Raise the head of my bed"
10. "I need my family at my bedside"

Picture board: Feasibility of communication using the BCI device will be evaluated using a picture board with illustrative icons representing the 10 needs/ complaints above as the standard for comparison and to determine the accuracy of selection of the appropriate icon. The icons and phrases on the picture board will be identical to the icons and phrases on the BCI device

SPECIFIC AIM 1:

To demonstrate the feasibility of using a Steady State Visual Evoked Potential (SSVEP) based Brain Computer Interface (BCI) device to facilitate communication of common patient needs in alert mechanically ventilated patients in the Intensive Care Unit (ICU).

Hypothesis 1: At least 80% of alert mechanically ventilated patients will be able to accurately select the illustrative icon on the brain computer interface representing the physical or emotional need self-identified by the patient as being the most common trigger for communication with the bedside nurse during their admission.

Orientation to BCI and picture board: The patient will initially be familiarized with both the picture board and the BCI device. Instruction on use of the BCI device will include demonstration of the UI, explanation of the icons on the UI and the mechanism of selection of an icon, through focused visual attention.

Selection of need/ complaint: Immediately following orientation, testing for accuracy of the BCI device will be performed. Testing for accuracy will be performed a single time for each patient, using the most important need/ complaint for that patient. The patient will be asked to identify on the BCI UI the specific need or complaint as being the most common reason to request the assistance of the bedside nurse during their admission, among the 10 patient need/ complaint options provided. Selection of "None of the above/ Other" will be permitted, however, the patient will be specifically instructed in advance to select the need/ complaint most applicable to their situation among the 10 choices provided. The patient will then be asked to select the SAME need/ complaint on the picture board using finger contact.

SPECIFIC AIM 2:

Specific Aim 2: To determine patient, family and bedside nurse satisfaction with communication using the BCI device and elicit open-ended feedback to guide future device improvements.

Hypothesis 2: At least 70% of patients will "agree" or "strongly agree" with the statement "The Brain computer interface device allowed me to communicate my needs to the bedside nurse adequately".

Immediately following evaluation of accuracy described under Specific Aim 1, the investigators will evaluate patient, family and bedside nurse satisfaction following bedside use of the device as the primary communication tool for 2 hours a day for 3 consecutive days. A delirium screen using CAM-ICU and a brief neurological examination to confirm the patient's ability to effectively use the BCI device and picture board will be performed prior to use of the device or picture board on subsequent days (days 2 and 3).

At the end of the 3 days, the patient, any family members present and each nurse who participated in testing will be provided the short questionnaires. The patient questionnaire with options will be read out to the patient.

Statistical Analysis:

The proportion of patients who pass Step 2 of screening who then also pass Step 3 will be calculated with exact binomial 95% confidence intervals. A proportion of at least 70% passing Step 3 of screening will be the initial threshold for feasibility, based on clinical estimates of value. The median time, with interquartile range, required for orientation to the BCI device and to the picture board will be calculated, and comparison performed using the Mann Whitney U-test. The proportion of patients who select the same icon on the BCI UI and the picture board will be calculated, with exact binomial 95% confidence intervals. In determining the accuracy of using the BCI device, a binomial analysis including multiple studies of BCI estimated the chance level at 63% (α = 0.05, 60 trials). Based also on a clinical estimate of what would be a minimum useful level of accuracy for a communication device, the threshold for accuracy in our study will be at least 80% of patients demonstrating concordance between selection of their most important need/ complaint on the BCI device and the picture board. Descriptive statistics will be used to for proportions of patients selecting responses to each of the satisfaction questions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an Intensive Care Unit and on mechanical ventilation for at least 24 hours
* Age 18 years or older
* Able to briskly follow commands
* Unimpaired use of at least one upper limb

Exclusion Criteria:

* Ongoing respiratory distress, severe pain or other source of obvious discomfort requiring immediate medical or nursing attention
* Severe hemodynamic instability with ongoing need for vasopressor titration or resuscitation
* Known impairment of vision, other than error of refraction with corrective lenses present
* Inability to tolerate interruption of sedation
* Inability to communicate fluently in English
* Need for ongoing EEG monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
BCI device accuracy | Immediately following enrollment
  Accurate selection of the illustrative icon on the brain computer interface representing the physical or emotional need self-identified by the patient as being the most common trigger for communication with the bedside nurse during their admission.

SECONDARY OUTCOMES:
Satisfaction survey | At the end of 3 days of using BCI device
  Selection by patients or family of "agree" or "strongly agree" with the statement "The Brain computer interface device allowed me to communicate my needs to the bedside nurse adequately".

CONTACTS AND LOCATIONS:
Overall Officials: Omid Dehzanghi, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Happ MB, Garrett K, Thomas DD, Tate J, George E, Houze M, Radtke J, Sereika S. Nurse-patient communication interactions in the intensive care unit. Am J Crit Care. 2011 Mar;20(2):e28-40. doi: 10.4037/ajcc2011433. PMID 21362711
- [Background] Johnson MM, Sexton DL. Distress during mechanical ventilation: patients' perceptions. Crit Care Nurse. 1990 Jul-Aug;10(7):48-57. No abstract available. PMID 2403412
- [Background] Carroll SM. Nonvocal ventilated patients perceptions of being understood. West J Nurs Res. 2004 Feb;26(1):85-103; discussion 104-12. doi: 10.1177/0193945903259462. PMID 14984652
- [Background] Baker C, Melby V. An investigation into the attitudes and practices of intensive care nurses towards verbal communication with unconscious patients. J Clin Nurs. 1996 May;5(3):185-92. doi: 10.1111/j.1365-2702.1996.tb00248.x. PMID 8705084
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Miglietta MA, Bochicchio G, Scalea TM. Computer-assisted communication for critically ill patients: a pilot study. J Trauma. 2004 Sep;57(3):488-93. doi: 10.1097/01.ta.0000141025.67192.d9. PMID 15454792
- [Background] Maringelli F, Brienza N, Scorrano F, Grasso F, Gregoretti C. Gaze-controlled, computer-assisted communication in Intensive Care Unit: "speaking through the eyes". Minerva Anestesiol. 2013 Feb;79(2):165-75. Epub 2012 Nov 22. PMID 23174919
- [Background] Smith E, Delargy M. Locked-in syndrome. BMJ. 2005 Feb 19;330(7488):406-9. doi: 10.1136/bmj.330.7488.406. No abstract available. PMID 15718541
- [Background] Daly JJ, Huggins JE. Brain-computer interface: current and emerging rehabilitation applications. Arch Phys Med Rehabil. 2015 Mar;96(3 Suppl):S1-7. doi: 10.1016/j.apmr.2015.01.007. PMID 25721542
- [Background] Chaudhary U, Birbaumer N, Curado MR. Brain-machine interface (BMI) in paralysis. Ann Phys Rehabil Med. 2015 Feb;58(1):9-13. doi: 10.1016/j.rehab.2014.11.002. Epub 2015 Jan 8. PMID 25623294
- [Background] Nijboer F, Sellers EW, Mellinger J, Jordan MA, Matuz T, Furdea A, Halder S, Mochty U, Krusienski DJ, Vaughan TM, Wolpaw JR, Birbaumer N, Kubler A. A P300-based brain-computer interface for people with amyotrophic lateral sclerosis. Clin Neurophysiol. 2008 Aug;119(8):1909-1916. doi: 10.1016/j.clinph.2008.03.034. Epub 2008 Jun 20. PMID 18571984
- [Background] Sellers EW, Ryan DB, Hauser CK. Noninvasive brain-computer interface enables communication after brainstem stroke. Sci Transl Med. 2014 Oct 8;6(257):257re7. doi: 10.1126/scitranslmed.3007801. PMID 25298323
- [Background] Marchetti M, Priftis K. Brain-computer interfaces in amyotrophic lateral sclerosis: A metanalysis. Clin Neurophysiol. 2015 Jun;126(6):1255-1263. doi: 10.1016/j.clinph.2014.09.017. Epub 2014 Oct 2. PMID 25449558
- [Background] Lesenfants D, Habbal D, Lugo Z, Lebeau M, Horki P, Amico E, Pokorny C, Gomez F, Soddu A, Muller-Putz G, Laureys S, Noirhomme Q. An independent SSVEP-based brain-computer interface in locked-in syndrome. J Neural Eng. 2014 Jun;11(3):035002. doi: 10.1088/1741-2560/11/3/035002. Epub 2014 May 19. PMID 24838215
- [Background] Muller-Putz GR, Scherer R, Brauneis C, Pfurtscheller G. Steady-state visual evoked potential (SSVEP)-based communication: impact of harmonic frequency components. J Neural Eng. 2005 Dec;2(4):123-30. doi: 10.1088/1741-2560/2/4/008. Epub 2005 Oct 25. PMID 16317236
- [Background] Herrmann CS. Human EEG responses to 1-100 Hz flicker: resonance phenomena in visual cortex and their potential correlation to cognitive phenomena. Exp Brain Res. 2001 Apr;137(3-4):346-53. doi: 10.1007/s002210100682. PMID 11355381
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Brunner P, Bianchi L, Guger C, Cincotti F, Schalk G. Current trends in hardware and software for brain-computer interfaces (BCIs). J Neural Eng. 2011 Apr;8(2):025001. doi: 10.1088/1741-2560/8/2/025001. Epub 2011 Mar 24. PMID 21436536
- See also: A practical VEP-based brain-computer interface — http://sccn.ucsd.edu/~yijun/pdfs/TNSRE06.pdf
- See also: BCIBench: A Benchmarking Suite for EEG-based Brain Computer Interface, ODES-11 2014 Workshop on Optimizations for DSP and Embedded Systems, February 15, 2014, Orlando, FL — http://odes-workshop.weebly.com/
- See also: A Novel Stimulation for Multi-Class SSVEP-Based Brain-Computer Interface Using Patterns of Time-Varying Frequencies, International Conference of the IEEE Engineering in Medicine and Biology Society (EMBC), August 26-30, 2014, Chicago, IL — http://jafari.tamu.edu/wp-content/uploads/2015/12/Omid_EMBC14.pdf
- See also: Frequency recognition based on canonical correlation analysis for SSVEP-based BCIs — http://ieeexplore.ieee.org/stamp/stamp.jsp?tp=&arnumber=4203016